CLINICAL TRIAL: NCT07145788
Title: The Effect of Physiotherapy Integrated With Yoga and Mindfulness on Disability in Individuals With Fibromyalgia: A Single-Blind Randomized Controlled Trial (PhYoMind)
Brief Title: The Effect of Physiotherapy Integrated With Yoga and Mindfulness on Disability in Individuals With Fibromyalgia
Acronym: PhYoMind
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260/2025BO2; 1059B142400174 (Other Grant/Funding Number: TÜBITAK)
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Fibromyalgia (FM)
Keywords: Mind-Body Intervention; Fibromyalgia; chronic pain; pain management; post-isometric relaxation; proprioceptive neuromuscular facilitation; physical therapy techniques
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Agnosia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Data analysis will also be conducted blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PhYoMind Intervention Group (Experimental): Physiotherapy techniques + yoga + mindfulness + home exercise
  Interventions: Other: PhYoMind
- Home Exercise Group (Active Comparator): Only Home Exercise (walking + strenghtening + streching)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: PhYoMind — This integrative intervention method includes some specific physiotherapy techniques, ( e. g. self proprioceptive neuromuscular facilitation, self nerve gliding, self mobility, post isometric relaxation techniques) yoga postures, left nostril breathing, humming bee breathing, mindfulness practices and home exercises. Each session will be 75 minutes and focus on different parts of the body and yoga postures will be selected according to these focused areas. For each week, a specific body area will be chosen as the focus. For example, the first week will focus on the hip area and lower extremities, the second week on the upper body and upper extremities, the third week on the core and anterior line of the body, and the fourth week on the back and posterior line of the body and this sequence will continue through the eighth week. In addition to these sessions, participants in this group will also apply home exercises (aerobic+strenghtening+streching) twice a week, 60 minutes per practice.
  Arms: PhYoMind Intervention Group
Other: Exercise — The control group will receive only home exercises twice a week. Big muscle groups strengthening and stretching exercises and walking planned for the patient will be given as home exercise. The walking exercise will last 30 minutes at a moderately fast pace, depending on the subject's adaptation. The strengthening exercises will last 15 minutes and will consist of 3 sets of 12 repetitions of exercises with body weight and light weights, generally targeting the back extensor muscles, core stabilization muscles, shoulder region muscles in the upper extremity and hip and knee joint muscles in the lower extremity. The stretching exercises will last 15 minutes and will include neck muscles, pectoralis major/minor, erector spina, hamstrings, quadriceps femoris muscles 1-2 times for 30 seconds each. Participants will be taught face to face with a brochure when they come for the first assessment and will be asked to do HE at home.
  Arms: Home Exercise Group

SUMMARY:
The current study investigates the effect of an integrative physiotherapy and mind-body programme called PhYoMind on disability in individuals with fibromyalgia (FM). Participants will be randomized to either the PhYoMind intervention, which combines specific physiotherapy techniques with yoga and mindfulness, or to a home-based exercise control group. The intervention lasts 8 weeks, with supervised and home sessions. The primary outcome is disability, with secondary outcomes including measures of central and autonomic nervous system function, pain, stress, fatigue, and sleep.

DETAILED DESCRIPTION:
FM is a chronic disorder characterized by widespread pain, fatigue, sleep disturbances, and cognitive-emotional difficulties. Despite its high prevalence, treatment options remain limited and often focus on symptom management rather than addressing underlying physiological dysregulation. Emerging evidence implicates abnormalities in the central nervous system (CNS) and autonomic nervous system (ANS), along with neurochemical imbalances, in the development and persistence of FM symptoms.

Although physiotherapy and mind-body practices such as yoga and mindfulness have individually shown benefits for fibromyalgia symptoms, there is a lack of research on combined interventions integrating these therapies.

The present randomized controlled trial investigates the effects of PhYoMind, a novel integrative program combining physiotherapy techniques - such as Proprioceptive Neuromuscular Facilitation (PNF), Nerve Gliding Exercises (NGE), Mobility Exercises (ME), and Post-Isometric Relaxation (PIR) - with yoga and mindfulness practices. The intervention aims to improve disability and address multiple symptoms in people with FM through an integrated approach.

Participants will be randomly assigned to receive either the PhYoMind program or a home-based stretching, strengthening, and aerobic exercise regimen over 8 weeks. Two supervised sessions per week will be complemented by prescribed home exercises. Outcomes will be assessed at baseline (Week 0) and immediately after post-intervention (Week 8), including disability (primary outcome), as well as pain, stress, fatigue, sleep quality, central nervous system function and autonomic function via heart rate variability.

This study will contribute valuable evidence regarding the potential benefits of an integrative physiotherapy and mind-body approach in managing fibromyalgia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of clinically diagnosed fibromyalgia according to the American College of Rheumatology

Exclusion Criteria:

* Other important causes of pain other than FM
* If participants have hypertension; in case of changes in antihypertensive medication during the study
* Severe osteoarthritis that affects activities of daily living
* Severe somatic or psychiatric disorders
* Receiving another physiotherapy and/or physical exercise treatment concurrently with this study
* Not having sufficient cognitive level or not being able to participate in the sessions.
* Participants must either be on a stable treatment for fibromyalgia or not receiving any treatment, with no intention to alter their treatment plan during the study period. Those who do not meet this criterion will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Disability, Fibromyalgia Impact Questionnaire (FIQ) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  The FIQ is a valid and reliable questionnaire with a total score range of 0-100 measuring overall disease severity, pain severity, physical functioning, work difficulties, morning fatigue, depression, anxiety, and general well-being rated by individuals with fibromyalgia. Higher scores indicate a greater impact of symptoms.

SECONDARY OUTCOMES:
Central Nervous System Assessment, Central Sensitization Inventory (CSI) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  This scale, which has a scoring system ranging from 0 to 100, consists of 25 items with a 5-point Likert type question, each of which is evaluated between 0 and 4 points. A total score of 40 and above is shown as a clinically significant cut-off value.
Autonomic Nervous System Assessment, Heart Rate Variability (HRV) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  Changes in the autonomic nervous system will be recorded by measuring heart rate variability. Heart Rate Variability (HRV) will be measured and recorded with a Polar H10 (Polar Electro UK Ltd., Warwick, UK) chest strap using the validated Elite HRV mobile application.
Current Pain Perception, The Visual Analog Scale (VAS) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  The Visual Analog Scale (VAS) scale, a widely used and valid and reliable scale, will be used to rate the pain intensity of the participants. The scale consists of a 10 cm long line, 0 "no pain"; 10 would represent "worst possible pain".
Fatique Assessment, The 20-item Multidimensional Fatigue Index (MFI) | At enrollment (Week 0) and after 8 weeks of intervention (Week 8)
  To measure the severity of fatigue in participants with fibromyalgia, the 20-item Multidimensional Fatigue Index (MFI), covering various aspects of fatigue (five subscales; general fatigue, physical fatigue, mental fatigue, decreased motivation, decreased activity) will be applied. Higher score indicates more severe fatigue.
Sleep Assessment, Pittsburgh Sleep Quality Index (PSQI) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  The questionnaire consists of 19 questions grouped into seven component scores, each with a range of 0-3, including specific sleep-related problems such as average sleep duration, sleep latency, and daytime sleepiness. An overall PSQI score (range 0 to 21) is calculated. Higher scores indicate poorer sleep quality.
Stress Assessment, Perceived Stress Scale (PSS) | At baseline (Week 0) and after 8 weeks of intervention (Week 8)
  This 10-item self-report scale is Likert-type and has a 5-point scoring system ranging from "never" to "very often". Higher scores were associated with higher perceived severity of stress.

OTHER OUTCOMES:
Demographic Data | At Baseline (Week 0)
  Participants' age (years), gender (male/female/other), years with FM diagnosis, medications, marital status, educational level, employment status, smoking status, and alcohol use will be measured.
weight (kg) | At Baseline (Week 0)
  Demographic Data
height (m) | At Baseline (Week 0)
  Demographic Data

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, Prof. Dr., Principal Investigator — Institute of General Practice and Interprofessional Care, University Hospital Tübingen, Tübingen, Germany
Locations (1):
- Bosch Health Campus, Stuttgart, Auerbachstraße 112, Germany

IPD SHARING:
Plan to Share IPD: No
Due to concerns regarding participant confidentiality and data privacy, as well as compliance with ethical approval and consent agreements, individual participant data will not be shared beyond the study team.